CLINICAL TRIAL: NCT00673699
Title: Observational: Studies in Human Beings Health Outcomes
Brief Title: The Role of Narrow-Band Imaging Endoscopy in Diagnosing Gastric Intestinal Metaplasia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Zvi Fireman MD, Head ,Gastroenterology Dept., Zvi Fireman MD, Gastroenterology Dept. Hillel Yaffe Med Ctr
Other Study IDs: HY-07/2008
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Dyspepsia
Keywords: NBI; gastroscopy; biopsy; intestinal metaplasia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gastric mucosal biopsy during upper gastrointestinal endoscopy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- A: Seventy dyspeptic consecutive patients that going upper gastrointestinal endoscopy
  Interventions: Procedure: Gastric mucosal biopsy

INTERVENTIONS:
Procedure: Gastric mucosal biopsy — Using upper gastrointestinal endoscopy with targeting biopsy in patients with dyspepsia
  Other Names: patients ith dyspepsia

SUMMARY:
The purpose of this study is to determine if endoscope with NBI(narrow banding imaging)can detect intestinal metaplasia( consider pre malignant condition) and use a targeting biopsy in case of suspected intestinal metaplasia

DETAILED DESCRIPTION:
To detect intestinal metaplasia which consider pre malignant condition and use a targeting biopsy in case of suspected intestinal metaplasia which allowed us to better follow-up those patients.

ELIGIBILITY:
Inclusion Criteria:

* Dyspepsia

Exclusion Criteria:

* Pregnancy,
* Upper gastrointestinal bleeding,
* Previous gastric operation,
* Known gastric malignancy'
* Non cooperative patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hundred consecutive dyspeptic patients
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
To determine if endoscope with NBI can detect intestinal metaplasia | In one week (the time from biopsy till the histology assement)

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Fireman, MD, Principal Investigator — Hillel Yaffe Med Ctr
Locations (1):
- Hillel Yaffe Med Ctr, Hadera, Israel

REFERENCES:
- [Background] Hirata M, Tanaka S, Oka S, Kaneko I, Yoshida S, Yoshihara M, Chayama K. Evaluation of microvessels in colorectal tumors by narrow band imaging magnification. Gastrointest Endosc. 2007 Nov;66(5):945-52. doi: 10.1016/j.gie.2007.05.053. PMID 17963882